CLINICAL TRIAL: NCT05258149
Title: Comparison of a Silicone Hydrogel Daily Disposable Multifocal Contact Lens to a Marketed Product
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CR-6479
Record Dates: First submitted 2022-02-17; First posted 2022-02-28 (Actual); Results first posted 2023-05-19 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-04

CONDITIONS: Visual Acuity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- TEST/CONTROL/CONTROL (Experimental): Eligible subjects will be randomized into the sequence TEST/CONTROL/CONTROL.
  Interventions: Device: JJVC Investigational Multifocal Contact Lenses; Device: Dailies Total 1® Multifocal Contact Lenses
- CONTROL/TEST/TEST (Experimental): Eligible subjects will be randomized into the sequence CONTROL/TEST/TEST
  Interventions: Device: JJVC Investigational Multifocal Contact Lenses; Device: Dailies Total 1® Multifocal Contact Lenses

INTERVENTIONS:
Device: JJVC Investigational Multifocal Contact Lenses — TEST
Device: Dailies Total 1® Multifocal Contact Lenses — CONTROL

SUMMARY:
This is a single-masked, 2×3 crossover, randomized-controlled, dispensing clinical trial to evaluate overall quality of vision.

ELIGIBILITY:
Inclusion Criteria:

* Potential subjects must satisfy all of the following criteria to be enrolled in the study

  1. Read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
  2. Appear able and willing to adhere to the instructions set forth in this clinical protocol.
  3. Be at least 40 years of age and not greater than 70 years of age at the time of consent.
  4. Own a wearable pair of spectacles if required for their distance vision.
  5. Be an adapted soft contact lens wearer in both eyes (i.e. worn lenses a minimum of 2 days per week for at least 6 hours per wear day, for 1 month or more duration).
  6. Either already be wearing a presbyopic contact lens correction (e.g., reading spectacles over contact lenses, multifocal or monovision contact lenses, etc.) or if not respond positively to at least one symptom on the "Presbyopic Symptoms Questionnaire" (Appendix D).
  7. The subject's distance spherical equivalent refraction (vertex corrected if ≥-4.25 D) must be in the range of -1.25 D to -5.75 D or +0.75 D to +3.25 D in each eye.
  8. The subject's refractive cylinder must be ≤0.75 D in each eye.
  9. The subject's ADD power must be in the range of +0.75 D to +2.50 D.
  10. The subject must have distance best corrected visual acuity of 20/20-3 or better in each eye.

      Exclusion Criteria:
* Potential subjects who meet any of the following criteria will be excluded from participating in the study:

The subject must not:

1. Be currently pregnant or lactating.
2. Have any active or ongoing ocular or systemic allergies that may interfere with contact lens wear.
3. Have any active or ongoing systemic disease, autoimmune disease, or use of medication, which may interfere with contact lens wear. This may include, but not be limited to, diabetes, hyperthyroidism, Sjögren's syndrome, xerophthalmia, acne rosacea, Stevens-Johnson syndrome, and immunosuppressive diseases or any infectious diseases (e.g. hepatitis, tuberculosis).
4. Have any previous, or planned, ocular or intraocular surgery (e.g. radial keratotomy, PRK, LASIK, lid procedures, dacryocystorhinostomy, peripheral iridotomy/iridectomy, cataract surgery, retinal surgery, etc.).
5. Have a history of amblyopia, strabismus or binocular vision abnormality.
6. Use of any of the following medications within 1 week prior to enrollment: oral retinoid, oral tetracyclines, anticholinergics, oral phenothiazines, oral/inhaled corticosteroids. See section 9.1 for further examples.
7. Use of any ocular medication, with the exception of rewetting drops.
8. Have a history of herpetic keratitis.
9. Have a history of irregular cornea.
10. Have a history of pathological dry eye.
11. Have Participated in any contact lens or lens care product clinical trial within 30 days prior to study enrollment.
12. Be an employee or immediate family member of an employee of clinical site (e.g., Investigator, Coordinator, Technician).
13. Have any known hypersensitivity or allergic reaction to non-preserved rewetting drop solutions or sodium fluorescein.
14. Have clinically significant (Grade 2 or greater) corneal edema, corneal vascularization, corneal staining, tarsal abnormalities or bulbar injection, or any other corneal or ocular abnormalities which would contraindicate contact lens wear.
15. Have any current ocular infection or inflammation.
16. Have any current ocular abnormality that may interfere with contact lens wear.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2022-02-18 (Actual); Primary Completion 2022-04-29 (Actual); Study Completion 2022-04-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Vision Care, Inc. Clinical Trial, Study Director — Johnson & Johnson Vision Care, Inc.
Locations (12):
- United States (12):
  - Vue Optical Boutique, Jacksonville, Florida
  - Stam & Associates Eye Care, Jacksonville, Florida
  - Sabal Eye Care, Longwood, Florida
  - Maitland Vision Center, Maitland, Florida
  - VisualEyes, Roswell, Georgia
  - Complete Eye Care of Medina, Medina, Minnesota
  - Spectrum Eyecare, Jamestown, New York
  - Eye Associates of New York, Manhattan, New York
  - Sacco Eye Group, Vestal, New York
  - ProCare Vision Centers, Granville, Ohio
  - Tyler Eye Associates, Tyler, Texas
  - Botetourt Eyecare, LLC, Salem, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 143 subjects were enrolled in this study. Of those enrolled, all 143 subjects were dispensed at least one study lens. Of those dispensed, 138 subjects completed the study while 5 subjects were discontinued.
Groups:
- Senofilcon A C3/Delefilcon A/Delefilcon A: Subjects in this sequence were randomized to receive the senofilcon A C3 lens during the first period and the delefilcon A lens during the second and third periods.
- Delefilcon A/Senofilcon A C3/Senofilcon A C3: Subjects in this sequence were randomized to receive the delefilcon A lens during the first period and the senofilcon A C3 lens during the second and third periods.
Period: Period 1
Arm/Group | Senofilcon A C3/Delefilcon A/Delefilcon A | Delefilcon A/Senofilcon A C3/Senofilcon A C3
Started | 70 | 73
Completed | 69 | 72
Not Completed | 1 | 1
Not completed — Protocol Deviation | 1 | 0
Not completed — Adverse Event | 0 | 1
Period: Period 2
Arm/Group | Senofilcon A C3/Delefilcon A/Delefilcon A | Delefilcon A/Senofilcon A C3/Senofilcon A C3
Started | 69 | 72
Completed | 68 | 71
Not Completed | 1 | 1
Not completed — Unsatisfactory Visual Response due to Test Article | 1 | 0
Not completed — Subject No Longer Meets Eligibility Criteria | 0 | 1
Period: Period 3
Arm/Group | Senofilcon A C3/Delefilcon A/Delefilcon A | Delefilcon A/Senofilcon A C3/Senofilcon A C3
Started | 68 | 71
Completed | 68 | 70
Not Completed | 0 | 1
Not completed — Subject Was Not Returning for More Than A Week | 0 | 1

BASELINE CHARACTERISTICS:
Population: All subjects dispensed at least one study lens.
Groups:
- Hyperopes: Subjects were classified as Hyperopic if the distance spherical equivalent refraction was in the range of +0.75 D to +3.25 D.
- Myopes: Subjects were classified as Myopic if the distance spherical equivalent refraction was in the range of -5.75 D to -1.25 D.
- Total: Total of all reporting groups
Arm/Group | Hyperopes | Myopes | Total
Number analyzed (Participants) | 56 | 87 | 143
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.3 (6.41) | 49.0 (5.84) | 52.3 (7.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 69 | 114
  Male | 11 | 18 | 29
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 2 | 4 | 6
  Black or African American | 1 | 11 | 12
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  White | 51 | 72 | 123
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 56 | 87 | 143

OUTCOME MEASURES:

1. Primary Outcome: Clarity of Vision in Dim or Low Lighting
Description: Clarity of vision in dim or low lighting was assessed at the 1-week follow-up during each study period using the individual item: Clarity of vision in dim or low lighting conditions. This item used a 5-point like-rt scale of (1=Excellent, 2=Very good, 3=Good, 4=Fair and 5=Poor). Results were presented as the percentage of subjects' responses in each category by lens. For analysis and summary purposes three categories were used (T2B-Excellent and Very Good, Middle Box-Good and B2B-Fair and Poor). The 1-week follow-up from each study period (1, 2 and 3) were all included in the summary.
Time Frame: 1-Week Follow-up
Population: All dispensed subjects regardless of deviation from protocol and completion status.
Measure: Number; unit: Percent
Units Other Than Participants: Observations
Groups:
- Senofilcon A C3: Subjects that wore the senofilcon A C3 lens during any of the three study periods.
- Delefilcon A: Subjects that wore the delefilcon A lens during any of the three study periods.
Arm/Group | Senofilcon A C3 | Delefilcon A
Number analyzed (Participants) | 143 | 143
Number analyzed (Observations) | 210 | 208
Percent
  Excellent or Very Good | 54.3 | 43.3
  Good | 33.3 | 36.1
  Fair or Poor | 12.4 | 20.6
Statistical Analysis 1: Comparison: Senofilcon A C3 vs Delefilcon A; Test type: Superiority — A superiority margin of 1 was used; Generalized Linear Mixed Model; Kenward and Roger Method was used for the denominator degrees of freedom; Odds Ratio (OR) = 1.65, 95% CI 2-sided [1.10 to 2.46] — Odds Ratio was calculated as senofilcon A C3 over delefilcon A

2. Primary Outcome: Clarity of Vision When Reading in Dim Light
Description: Clarity of vision when reading in dim light was assessed at the 1-week follow-up during each study period using the individual item: Clarity of vision when reading in dim light(e.g., menu or bill in a restaurant). This item used a 5-point like-rt scale of (1=Excellent, 2=Very good, 3=Good, 4=Fair and 5=Poor). Results were presented as the percentage of subjects' responses in each category by lens. For analysis and summary purposes three categories were used (T2B-Excellent and Very Good, Middle Box-Good and B2B-Fair and Poor). The 1-week follow-up from each study period (1, 2 and 3) were all included in the summary.
Time Frame: 1-Week Follow-up
Population: All dispensed subjects regardless of deviation from protocol and completion status.
Measure: Number; unit: Percent
Units Other Than Participants: Observations
Arm/Group | Senofilcon A C3 | Delefilcon A
Number analyzed (Participants) | 143 | 143
Number analyzed (Observations) | 210 | 208
Percent
  Excellent or Very Good | 46.2 | 32.2
  Good | 32.4 | 34.1
  Fair or Poor | 21.4 | 33.6
Statistical Analysis 1: Comparison: Senofilcon A C3 vs Delefilcon A; Test type: Superiority — A superiority margin of 1 was used; Generalized Linear Mixed Model; Kenward and Roger Method was used for the denominator degrees of freedom; Odds Ratio (OR) = 1.88, 95% CI 2-sided [1.27 to 2.79] — Odds Ratio was calculated as senofilcon A C3 over delefilcon A

3. Secondary Outcome: Clarity of Distance Vision
Description: Clarity of Distance vision was assessed at the 1-week follow-up during each study period using the individual item: Clarity of distance vision (i.e., looking at things that are more than 5 feet away, such as street signs). This item used a 5-point like-rt scale of (1=Excellent, 2=Very good, 3=Good, 4=Fair and 5=Poor). Results were presented as the percentage of subjects' responses in each category by lens. For analysis and summary purposes three categories were used (T2B- Excellent and Very Good, Middle Box-Good and B2B- Fair and Poor). The 1-week follow-up from each study period (1, 2 and 3) were all included in the summary.
Time Frame: 1-Week Follow-up
Population: All dispensed subjects regardless of deviation from protocol and completion status.
Measure: Number; unit: Percent
Units Other Than Participants: Observations
Arm/Group | Senofilcon A C3 | Delefilcon A
Number analyzed (Participants) | 143 | 143
Number analyzed (Observations) | 210 | 208
Percent
  Excellent or Very Good | 70.4 | 74.1
  Good | 21.9 | 21.6
  Fair or Poor | 7.7 | 4.3
Statistical Analysis 1: Comparison: Senofilcon A C3 vs Delefilcon A; Test type: Non-Inferiority — A Non-Inferiority margin of 10% was used; Generalized Linear Mixed Model; Kenward and Roger Method was used for the denominator degrees of freedom; Odds Ratio (OR) = 0.74, 98.33% CI 2-sided [0.42 to 1.30] — Odds Ratio was calculated as senofilcon A C3 over delefilcon A; confidence intervals were adjusted using 98.33% per each secondary endpoint

4. Secondary Outcome: Clarity of Intermediate Vision
Description: Clarity of Intermediate vision was assessed at the 1-week follow-up during each study period using the individual item: Clarity of intermediate vision (i.e., looking at things 2-3 feet away, such as your computer screen). This item used a 5-point like-rt scale of (1=Excellent, 2=Very good, 3=Good, 4=Fair and 5=Poor). Results were presented as the percentage of subjects' responses in each category by lens. For analysis and summary purposes three categories were used (T2B-Excellent and Very Good, Middle Box-Good and B2B-Fair and Poor). The 1-week follow-up from each study period (1, 2 and 3) were all included in the summary.
Time Frame: 1-Week Follow-up
Population: All dispensed subjects regardless of deviation from protocol and completion status.
Measure: Number; unit: Percent
Units Other Than Participants: Observations
Arm/Group | Senofilcon A C3 | Delefilcon A
Number analyzed (Participants) | 143 | 143
Number analyzed (Observations) | 210 | 208
Percent
  Excellent or Very Good | 75.2 | 64.4
  Good | 21.0 | 27.9
  Fair or Poor | 3.8 | 7.7
Statistical Analysis 1: Comparison: Senofilcon A C3 vs Delefilcon A; Test type: Superiority — A superiority margin of 1 was used; Generalized Linear Mixed Model; Kenward and Roger Method was used for the denominator degrees of freedom; Odds Ratio (OR) = 1.58, 98.33% CI 2-sided [0.91 to 2.75] — Odds Ratio was calculated as senofilcon A C3 over delefilcon A; confidence intervals were adjusted using 98.33% per each secondary endpoint

5. Secondary Outcome: Clarity of Near Vision
Description: Clarity of Near vision was assessed at the 1-week follow-up during each study period using the individual item: Clarity of intermediate vision (i.e., looking at things close up, such as reading a book). This item used a 5-point like-rt scale of (1=Excellent, 2=Very good, 3=Good, 4=Fair and 5=Poor). Results were presented as the percentage of subjects' responses in each category by lens. For analysis and summary purposes three categories were used (T2B-Excellent and Very Good, Middle Box-Good and B2B-Fair and Poor). The 1-week follow-up from each study period (1, 2 and 3) were all included in the summary.
Time Frame: 1-Week Follow-up
Population: All dispensed subjects regardless of deviation from protocol and completion status.
Measure: Number; unit: Percent
Units Other Than Participants: Observations
Arm/Group | Senofilcon A C3 | Delefilcon A
Number analyzed (Participants) | 143 | 143
Number analyzed (Observations) | 210 | 208
Percent
  Excellent or Very Good | 52.3 | 38.0
  Good | 35.7 | 35.1
  Fair or Poor | 12 | 26.9
Statistical Analysis 1: Comparison: Senofilcon A C3 vs Delefilcon A; Test type: Superiority — A superiority margin of 1 was used; Generalized Linear Mixed Model; Kenward and Roger Method was used for the denominator degrees of freedom; Odds Ratio (OR) = 2.08, 98.33% CI 2-sided [1.24 to 3.50] — Odds Ratio was calculated as senofilcon A C3 over delefilcon A; confidence intervals were adjusted using 98.33% per each secondary endpoint

ADVERSE EVENTS:
Time Frame: Throughout the duration of the study; Approximately 17-21 days per subject.
Arm/Group | Senofilcon A C3 | Delefilcon A
All-Cause Mortality (participants affected / at risk) | 0/142 | 0/142
Serious Adverse Events (participants affected / at risk) | 0/142 | 0/142
Other Adverse Events (participants affected / at risk) | 0/142 | 0/142

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-15): https://cdn.clinicaltrials.gov/large-docs/49/NCT05258149/Prot_SAP_000.pdf